CLINICAL TRIAL: NCT03191409
Title: Interaction Research on Cognitive Impairment and Emotional Disorder in End-stage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xidian University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015YK15
Record Dates: First submitted 2016-06-22; First posted 2017-06-19 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: End-stage Kidney Disease; Brain Damage
Keywords: cognitive impairment; ESRD; functional MRI
MeSH Terms: conditions — Kidney Failure, Chronic; Brain Injuries; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Health adults with no evidence of brain lesions on conventional magnetic resonance imaging(MRI) and no neural developmental disorders.
- Patients Group: ESRD patients pre-hemodialysis will be collected.The following exclusion criteria were applied in this study: (a)history of drug or alcohol abuse, (b) brain lesions such as a tumor or stroke assessed on the basis of medical history, (c) history of or current psychiatric disorders, and (d) head motion more than 1.0 mm or 1.0°during magnetic resonance imaging. All patients completed laboratory tests to evaluate renal function,serum creatinine, and urea levels within the 12 hours before magnetic resonance imaging.

SUMMARY:
End stage renal disease (ESRD) is the last stage (stage 5) of chronic kidney disease (CKD). Abnormalities of cognitive function and high levels of depression or anxiety incidence are characteristic of hemodialysis patients. In this research project, the investigators subject in ESRD patients starting hemodialysis as the carrier. Based on the longitudinal research design, using multimodal neuroimaging data，combining with the interact relationship between changes of brain morphology, the dysfunction of resting-state and-task state with cognitive impairment and abnormal emotions.Establish brain structure-function change model associated with dialysis progression, Explore imaging markers of central and disease development characteristics in ESRD patients. the investigators attempt to clarify the core mechanism of kidney-brain axis damage, thus provide evidence for early cognitive-behavioral therapy to CKD patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years;
2. ESRD patients who will start hemodialysis
3. High quality MRI scan;
4. dextromanual

Exclusion Criteria:

1. Diabetes,Brain tumor,brain trauma
2. Neuropsychiatric disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ESRD patients before dialysis initiation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
change in cognitive function | Change from Baseline to 3 Months after dialysis
  Cognitive testing will be performed for assessment

SECONDARY OUTCOMES:
Change in brain MRI | Change from Baseline to 3 Months after dialysis
  Brain MRI will be performed before dialysis initiation and dialysis more than 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided